CLINICAL TRIAL: NCT00942123
Title: On the Role of Mitochondrial Dysfunction in the Pathogenesis of Metformin-associated Lactic Acidosis
Brief Title: Study On the Role of Mitochondrial Dysfunction in the Pathogenesis of Metformin-associated Lactic Acidosis
Status: Completed | Type: Observational
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Responsible Party: Sponsor
Other Study IDs: 2551
Record Dates: First submitted 2009-07-16; First posted 2009-07-20 (Estimated); Last update posted 2013-09-27 (Estimated); Status verified 2013-09

CONDITIONS: Lactic Acidosis; Metformin
MeSH Terms: conditions — Acidosis, Lactic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Metformin is the first line drug of choice for the treatment of type II diabetes. Lactic acidosis can develop as a side effect, especially when renal failure leads to drug accumulation. Lactic acidosis is usually attributed to an abnormal inhibition of hepatic lactate clearance.

Growing evidence suggest that metformin can dose-dependently inhibit hepatocyte mitochondrial function. Whether a similar effect occurs in extra-hepatic human tissues remains unknown.

The investigators hypothesize that mitochondrial dysfunction occurs during metformin intoxication even in tissues other than the liver, thus contributing to the development of lactic acidosis. The aim of this study is to investigate mitochondrial integrity in circulating platelets of patients with lactic acidosis due to metformin intoxication.

ELIGIBILITY:
Inclusion Criteria:

1. Lactic acidosis (pH < 7.35 or base deficit > 5 mmol/L and lactate > 5 mmol/L)
2. Metformin intoxication (serum drug level > 4 mcg/mL)
3. Absence of evidence of any other condition that could primarily explain the lactic acidosis

Exclusion Criteria:

1. Less than 18 years of age
2. Hemoglobin < 8 g/dL (10 g/dL if ischemic cardiac disease)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with lactic acidosis and metformin intoxication (as documented by drug serum measurement)
Sampling Method: Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2009-01; Primary Completion 2010-12 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Platelet mitochondrial respiratory chain enzyme activity | Within 48 hours from admission to ICU

CONTACTS AND LOCATIONS:
Locations (1):
- Ospedale Maggiore Policlinico, Milan, MI, Italy

REFERENCES:
- [Derived] Protti A, Lecchi A, Fortunato F, Artoni A, Greppi N, Vecchio S, Fagiolari G, Moggio M, Comi GP, Mistraletti G, Lanticina B, Faraldi L, Gattinoni L. Metformin overdose causes platelet mitochondrial dysfunction in humans. Crit Care. 2012 Oct 3;16(5):R180. doi: 10.1186/cc11663. PMID 23034133